CLINICAL TRIAL: NCT04337684
Title: Long Term Follow-Up and Collection of Historical Control Data on Menkes Disease Patients
Brief Title: Long Term Follow-up on Menkes Disease Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Cyprium Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CYP-002
Record Dates: First submitted 2020-04-01; First posted 2020-04-08 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Menkes Disease
MeSH Terms: conditions — Menkes Kinky Hair Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Historical Control
- Treated with Copper Histidinate
  Interventions: Drug: Long Term Follow-Up

INTERVENTIONS:
Drug: Long Term Follow-Up — Menkes disease is a form of inherited copper deficiency associated with neurodevelopmental delays and neurological problems. Copper Histidinate is being evaluated for efficacy and safety in patients with Menkes disease. The purpose of this protocol is to collect long term follow-up data.
  During the study, patients and/or parent/legal guardian will be contacted by the investigator by either telephone or an in-person visit to assess long term follow-up.
  Other Names: CUTX-101
  Groups: Treated with Copper Histidinate

SUMMARY:
This study will collect long term follow-up data regarding overall survival and neurological parameters from patients previously identified and/or enrolled in Protocols 09-CH-0059 and 90-CH0149 and Historical Control data on Menkes disease patients.

DETAILED DESCRIPTION:
Primary Objective:

1. To provide additional clinical and safety data on long term following administration of Copper Histidinate treatment in patients treated with Copper Histidinate under Protocols 09-CH-0059 and 90-CH0149 and untreated patients previously identified and/or enrolled in Protocol 09-CH-0059.
2. To provide additional Historical Control data on Menkes disease patients.

ELIGIBILITY:
Inclusion Criteria:

* The subject must have been previously identified and/or enrolled under Protocols 09-CH-0059 or 90-CH-0149; or An untreated Menkes disease patients for whom data collection is incomplete under Protocols 09-CH-0059 (Amendment M); or Other untreated Menkes disease patients.
* Must sign and date an informed consent form by parent or legal guardian for this study prior to any assessment being done in this study. If the patient is > 18 years of age, the patient must sign the informed consent.
* Male or female, aged 0 to < 65 years of age.

Exclusion Criteria:

- Unwillingness/unable to participate in the study.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 1. Any subject previously identified and/or enrolled in either Protocols 09-CH-0059 or 90-CH-0149.
  2. Any new untreated Menkes disease patient born after 1999.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Long Term Follow-Up on Survival | 12/01/2019 - 12/31/2022
  The primary outcome measure will be overall survival.

CONTACTS AND LOCATIONS:
Locations (1):
- Cyprium Study Team, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided